CLINICAL TRIAL: NCT00003353
Title: A Phase II Study of High-Dose Melphalan With Hematopoietic Stem Cell Reconstitution for Patients With Primary Systemic Amyloidosis
Brief Title: High-Dose Melphalan Plus Peripheral Stem Cell Transplantation in Treating Patients With Primary Systemic Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066334; E-4A97
Record Dates: First submitted 1999-11-01; First posted 2004-09-13 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: primary systemic amyloidosis
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Immunoglobulin Light-chain Amyloidosis | interventions — Filgrastim; Melphalan; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: melphalan
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: High-dose chemotherapy may destroy the amyloid-producing cells in bone marrow. Peripheral stem cell transplantation

PURPOSE: Phase II trial to study the effectiveness of high dose melphalan plus peripheral stem cell transplantation in treating patients who have primary systemic amyloidosis.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the response rate and overall survival of patients with biopsy proven primary amyloidosis following treatment with myeloablative chemotherapy and hematopoietic stem cell reconstitution. II. Evaluate the toxicity of high dose melphalan in this patient population.

OUTLINE: Patients receive filgrastim (G-CSF) subcutaneously daily beginning on day 1 of the peripheral blood stem cell (PBSC) collection period and continuing until PBSC collection is completed. PBSC are collected beginning on day 5 of the collection period and continuing until the final target cell count is reached or for up to a maximum of 7 collections. If sufficient PBSCs are not harvested within a maximum of 7 collections, the patient is removed from the study. Within 30 days of PBSC collection, patients receive melphalan IV on day -1 of the infusion period and PBSC infusion on day 0. The infusion period continues until day 30. Patients receive G-CSF subcutaneously daily starting on day 1 and continuing until blood counts recover. Patients are followed every 3 months for 2 years, every 3 months for 3 additional years, and yearly thereafter.

PROJECTED ACCRUAL: A maximum of 33 patients will be accrued for this study over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed primary amyloidosis Must have presence of paraprotein in serum or urine determined by immunoelectrophoresis/immunofixation No primary amyloidosis manifested only by carpal tunnel syndrome or purpura No history of secondary, familial, or localized amyloidosis No evidence of overt multiple myeloma: Lytic bone disease or pathological fractures OR At least 30% plasma cells in bone marrow

PATIENT CHARACTERISTICS: Age: 18 to 70 Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute granulocyte count at least 1000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL Alkaline phosphatase no greater than 1000 u/L or less than 4 times upper limit of normal Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: Confirmed by echocardiogram: Ejection fraction at least 50% Interventricular septal thickness no greater than 15 mm No New York Heart Association classification II-IV Pulmonary: DLCO at least 50% FVC at least 60% FEV1 at least 55% Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No active infection No other malignancy within the past 5 years except surgically treated carcinoma in situ of the cervix, nonmelanoma skin cancer, or indolent prostate cancer No known sensitivity to E. coli derivatives

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior interferon allowed Chemotherapy: At least 4 weeks since prior melphalan Lifetime cumulative dose of melphalan no greater than 150 mg No greater than 2 prior courses of chemotherapy Endocrine therapy: Prior dexamethasone allowed Radiotherapy: Not specified Surgery: Not specified

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-11-16 (Actual); Primary Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morie A. Gertz, MD, Study Chair — Mayo Clinic
Locations (17):
- United States (17):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - New England Medical Center Hospital, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - University of Rochester Cancer Center, Rochester, New York
  - Ireland Cancer Center, Cleveland, Ohio
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin

REFERENCES:
- [Result] Gertz MA, Blood E, Vesole DH, Abonour R, Lazarus HM, Greipp PR. A multicenter phase 2 trial of stem cell transplantation for immunoglobulin light-chain amyloidosis (E4A97): an Eastern Cooperative Oncology Group Study. Bone Marrow Transplant. 2004 Jul;34(2):149-54. doi: 10.1038/sj.bmt.1704539. PMID 15156165